CLINICAL TRIAL: NCT06166771
Title: Safety and Effectiveness of the Alma System in Treating Primary Postpartum Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ResQ Medical Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-01-001-PR; ResQ Medical IL # 516181633 (Other: ResQ Medical Ltd.)
Record Dates: First submitted 2023-11-29; First posted 2023-12-12 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Hemorrhage (PPH); Postpartum Hemorrhage (Primary); PPH
Keywords: alma, pph, post partum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Woman who developed PPH after vaginal birth and first line therapies have been attempted and failed (Experimental): Group which Alma treatment was applied
  Interventions: Device: Alma system

INTERVENTIONS:
Device: Alma system — Subjects diagnosed with postpartum hemorrhage will receive the Alma System. This system comprises a soft silicone cylindrical device placed within the uterus. Gentle suction is applied, prompting the uterus to contract and reduce in size. This contraction compresses the blood vessels, halting the bleeding.
  Other Names: Vacuum induced heamorrhage control; Obstetric-gynecologic specialized manual instrument

SUMMARY:
Postpartum Hemorrhage (PPH) is an obstetric emergency that can occur up to 24 hours after vaginal birth or cesarean section.

In most cases, the uncontrolled bleeding is due to a lack of sufficient contraction of the uterus (hypotonia) and appears immediately after birth.

The purpose of this prospective, non-randomized, feasibility pilot study is to obtain information on the safety and effectiveness of an investigational new medical device - Alma System, that is intended to provide control and treatment of abnormal postpartum uterine bleeding or hemorrhage when conservative management is warranted.

DETAILED DESCRIPTION:
A prospective, non-randomized, feasibility pilot study that is intended to obtain information on the safety and effectiveness of the Alma System.

Study population: Women with vaginal deliveries in a hospital setting who failed first-line therapies for postpartum hemorrhage.

The main questions are:

1. Rate of device related SAEs up to six weeks following device treatment.
2. Rate of any observable damage to cervix, uterus or vagina during or immediately after device procedure.
3. Rate of occurrence of uterine inversion of folding during or immediately after device procedure.

Main tasks for participants:

* sign the informed Consent form and enrolment
* In case of PPH, treatment with Alma
* Participate in 2 follow-up visits After the treatment- 1st upon discharge and 2nd after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female, 18 years of age or older at time of consent.
2. Subject or her legally authorized representative is able to understand and provide consent to participate in the clinical investigation.
3. Subjects who present with an atonic uterus for at least 10 minutes after expulsion of placement with failure to obtain contraction and/or Subjects who have lost blood post-partum > = 500 ml and according to the Investigator's judgment, require an intervention.
4. Failed first-line intervention of uterotonics and uterine massage/bimanual uterine massage to stop bleeding.

Exclusion Criteria:

1. Subjects who do not provide informed consent to participate in the clinical investigation.
2. Subjects who deliver at a uterus size < 34 weeks.
3. Subjects who have lost greater than 1000 ml of blood.
4. Subjects who have abnormal PT, PTT and INR
5. Subjects who present with retained placenta, uterine lacerations, or for any other conditions outside of atonic post-partum hemorrhage.
6. PPH that the investigator determines to require more aggressive treatment, including any of the following:

   * Hysterectomy;
   * B-lynch suture;
   * Uterine artery embolization or ligation;
   * Hypogastric ligation.
   * Known uterine anomaly.
   * Ongoing intrauterine pregnancy.
7. Placental abnormality including any of the following:

   * Known placenta accreta;
   * Retained placenta with known risk factors for placenta accreta (e.g., history of prior uterine surgery, including prior c-section and placenta previa);
   * Retained placenta without easy manual removal.
8. Known uterine rupture.
9. Unresolved uterine inversion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Related SAEs | 6 weeks
  Rate of device related SAEs up to six weeks following device treatment.
Rate of Damage to Cervix, Uterus or Vagina | When removing the Alma System at the end of the procedure
  Rate of any observable damage to cervix, uterus or vagina during or immediately after device procedure
Rate of Occurrence of Uterine Inversion or Folding | When removing the Alma System at the end of the procedure
  Rate of occurrence of uterine inversion or folding during or immediately after device procedure

SECONDARY OUTCOMES:
User Feedback on Placement of Alma | When removing the Alma System at the end of the procedure
  Rate of positive user feedback on device placement trans-vaginally
User Feedback on Connection to Vacuum | When removing the Alma System at the end of the procedure
  Rate of positive user feedback on connection to vacuum and maintenance of desired negative pressure
Rate of Uterine Contraction | When removing the Alma System at the end of the procedure
  Rate of uterine contraction to a level that reduces or stops blood flow
Time to Visible Reduction in Blood Flow | When removing the Alma System at the end of the procedure
  Time from insertion and start of negative pressure to visible reduction in blood flow

CONTACTS AND LOCATIONS:
Locations (1):
- UNIVERSITY OF NAIROBI (UoN) COLLEGE OF HEALTH SCIENCES, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No